CLINICAL TRIAL: NCT00402545
Title: A Phase I Study of Cetuximab/Docetaxel(Taxotere)/Cisplatin/5-Fluorouracil (C-TPF) in Patients With Newly Diagnosed Locally Advanced Squamous Cell Carcinoma of the Head and Neck
Brief Title: C-TPF in Patients With Newly Diagnosed Locally Advanced Squamous Cell Carcinoma of the Head and Neck
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Brigham and Women's Hospital (Other); Bristol-Myers Squibb (Industry)
Responsible Party: Robert Haddad, MD, Dana-Farber Cancer Institute
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 06-128; CA225249
Record Dates: First submitted 2006-11-21; First posted 2006-11-22 (Estimated); Last update posted 2009-11-02 (Estimated); Status verified 2009-10

CONDITIONS: Head and Neck Neoplasms
Keywords: SCCHN; C-TPF; 5-FU; squamous cell carcinoma of the head and neck
MeSH Terms: conditions — Head and Neck Neoplasms; Squamous Cell Carcinoma of Head and Neck | interventions — Cetuximab; Docetaxel; Cisplatin; Fluorouracil

INTERVENTIONS:
Drug: Cetuximab — Given intravenously on days 1, 8 and 15 of each 21-day cycle for three cycles
Drug: Docetaxel — Given intravenously on day 1 of each 21-day cycle for 3 cycles
  Other Names: Taxotere
Drug: Cisplatin — Intravenously on day 1 of each 21-day cycle for 3 cycles
Drug: 5-Fluorouracil — Given by continuous infusion pump over a period of 96 hours(dosage wil vary depending upon when participant enrolls in trial)
  Other Names: 5-FU

SUMMARY:
The purpose of this research study is to determine the safest and most effective dose of 5-FU that can be given with docetaxel (Taxotere), Cisplatin and cetuximab to patients with newly diagnosed locally advanced squamous cell carcinoma of the head and neck. We will also be studying the toxicity of this regimen of 4 drugs and the tumor response.

DETAILED DESCRIPTION:
* After the screening tests confirm the participants eligibility, study treatment will begin.
* Prior to the start of study medication a port-a-cath will be inserted. This is done in the operating room and will require a separate consent form. During treatment a needle will be inserted into the port-a-cath through which the chemotherapy will be given. If the participant chooses not to have a port-a-cath, they will need to be hospitalized at Brigham and Women's Hospital to receive chemotherapy (approximately 5 days).
* Participants will receive three cycles of chemotherapy. Each cycle of treatment will last 21 days. On day 1 of each cycle, they will receive cetuximab intravenously for 2 hours, docetaxel (Taxotere) intravenously for 1 hour, cisplatin intravenously for 1 hour, and 5-FU over a period of 96 hours through an infusion pump. On days 8 and 15 of each cycle, participants will receive another dose of cetuximab intravenously for one hour.
* Not everyone who participates in this study will receive the same amount of 5-FU. A small group of participants will be given a certain dose of 5-FU through a continuous 4 day infusion. If they tolerate that well, the next group of people will receive a higher dose of 5-FU. This will continue until we can find the highest dose of the drug that can be given safely.
* Participants will be seen once a week in the clinic for a physical exam. At this time vital signs will be checked and participants will be asked general questions about their health and specific questions about any problems they might be experiencing. Blood tests will also be performed at this time.
* Within two weeks of completion of the third cycle of chemotherapy, participants will return to the clinic for evaluation. The following exams and procedures will be performed: Physical exam; blood tests; imaging of tumor (CT, MRI or PET); exam under anesthesia (EUA).
* Once the participant has completed all treatment, we would like to follow-up with them regarding the status of their cancer. Follow-up appointments will occur every 4-6 weeks for the first year, every 8-10 weeks up to the second year, every 3 months for the third year, and then every 6 months until the fifth year.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically proven squamous cell carcinoma of the head and neck.
* Primary tumor sites eligible: oral cavity, oropharynx, nasopharynx, hypopharynx, or larynx. Unknown primary SCC will also be eligible.
* Stage 3 or 4 disease without evidence of distant metastases verified by chest x-ray, abdominal ultrasound or CAT scan.
* At lease one uni- or bi-dimensionally measurable lesion by RECIST criteria.
* 18 years of age or older
* ECOG performance status of 0-1
* Adequate bone marrow, hepatic and renal functions as outlined in the protocol.

Exclusion Criteria:

* Pregnant or breast feeding women
* Previous or current malignancies at other sites, with the exception of adequately treated in situ carcinoma of the cervix, basal or squamous cell carcinoma of the skin or other cancer curatively treated by surgery and with no evidence of disease for at least 5 years.
* Symptomatic peripheral neuropathy greater or equal to grade 2
* Symptomatic altered hearing > grade 2 by CIT-CTC criteria
* Unstable cardiac disease despite treatment, myocardial infarction within 6 months
* History of significant neurologic or psychiatric disorders including dementia or seizures
* Active clinically significant uncontrolled infection
* Active peptic ulcer disease defined as unhealed or clinically active
* Hypercalcemia
* Active drug addiction, including alcohol, cocaine or intravenous drugs use
* Chronic Obstructive Pulmonary Disease
* Autoimmune disease requiring therapy, prior organ transplant, or HIV infection
* Interstitial lung disease
* Involuntary weight loss of more than 25% of their body weight in the 2 months preceding study entry
* Concurrent treatment with any other cancer drug
* Prior EGFR therapy
* Prior severe infusion reaction to antibody therapy
* Participation in an investigational trial within 30 days of study entry

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Estimated)
Dates: Start 2007-01; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Determine the maximum tolerated dose (MTD) of Docetaxel/Cisplatin/5-Fluorouracil (TPF) induction chemotherapy when combined with cetuximab in an induction chemotherapy setting for locally advanced squamous cell cancer of the head and neck. | 2 years

SECONDARY OUTCOMES:
To asses toxicity of this combination | 2 years
To determine the response rate in this patient population. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Robert I Haddad, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Dana-Farber Cancer Institute, Boston, Massachusetts, United States